CLINICAL TRIAL: NCT02445664
Title: Effect of a Tablet-administered Educational Video on Patients´ Knowledge on Osteoporosis and Treatment - a Randomized, Controlled Trial
Brief Title: Effect of a Tablet-administered Educational Video on Patients´ Knowledge on Osteoporosis and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kirsa Skov, Student, pharmacist, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OP_77
Record Dates: First submitted 2015-05-08; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Osteoporosis
Keywords: Patient education; Video intervention
MeSH Terms: conditions — Osteoporosis

ARMS (2):
- Video intervention (Experimental): A tablet-administered educational video (10 minutes duration).
  Interventions: Behavioral: Educational video
- Control (No Intervention): No intervention (no video)

INTERVENTIONS:
Behavioral: Educational video — Video: Information on osteoporosis and alendronate treatment.
  Arms: Video intervention

SUMMARY:
Osteoporosis is a highly prevalent disease in which non-adherence is a well-recognized problem. Non-adherence may be due to patients´ lack of knowledge, understanding, and involvement. In this study the investigators aimed to determine the effect of an educational video displayed on a tablet-device. The investigators hypothesized that an educational video would increase patients´ knowledge on osteoporosis and treatment at a two week follow up.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for at DXA scan at the osteoporosis clinic
* Currently on once-weekly alendronate treatment
* Informed consent

Exclusion Criteria:

* Patients that do not understand Danish
* Patients having hearing impairments (unable to hear the video)
* Patients having visual impairments (unable to watch the video)
* Patients diagnosed with dementia
* Patients unable to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in knowledge score | Baseline and 2-week follow up

SECONDARY OUTCOMES:
Change in "confidence to treatment" score, as indicated by participant response to questionnaire. | Baseline and 2-week follow up
  Measured on a scale from 1-10
Change in "satisfaction with the amount of information" score, as indicated by participant response to questionnaire. | Baseline and 2-week follow up
  Measured on a scale from 1-10
Change in "understandability of the information" score, as indicated by participants response to questionnaire. | Baseline and 2-week follow up
  Measured on a scale from 1-10